CLINICAL TRIAL: NCT07059091
Title: Clinical Trial of Omalizumab for Allergen Sensitized and Exposed Individuals With COPD (COPD-OMA)
Brief Title: Clinical Trial of Omalizumab for Allergen Sensitized and Exposed Individuals With COPD
Acronym: COPD-OMA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Genentech, Inc. (Industry); American Lung Association Asthma Clinical Research Centers (Other); American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00498976; 1U01AI177195 (NIH)
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Allergies
Keywords: lung disease; COPD; allergies
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypersensitivity; Lung Diseases | interventions — Omalizumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Multicenter phase II placebo-controlled, masked, randomized superiority clinical trial of omalizumab vs placebo in individuals with COPD having sensitization and exposure to indoor allergens.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participant and the study team (e.g., PI, study physician, coordinator), with the exception of an unblinded individual, will remain masked during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Omalizumab injection (Active Comparator): Active treatment is omalizumab injection, dosed using standardized weight and total IgE based table, as used for asthma treatment
  Interventions: Drug: Omalizumab (Xolair®)
- Placebo injection (Placebo Comparator): Placebo for omalizumab used in the study will be commercially packaged 0.9% Sodium Chloride Injection, USP (e.g., normal saline). The injection volumes of normal saline administered will be calculated based upon the volume of active omalizumab expected to be administered based upon weight and total IgE level.
  Interventions: Drug: Sodium Chloride (NaCl) 0.9 %

INTERVENTIONS:
Drug: Omalizumab (Xolair®) — The study drug (omalizumab or placebo) will be given as a subcutaneous injection, which means an injection into the fat layer just under the skin in your arm or leg. This is similar to an insulin injection and not as deep as a typical vaccine injection. After the injection, participants will be monitored for any side effects. The study team will determine the dose and how often the injection is given based on the participant's weight and blood test results. Injections will be either be given monthly, 12 doses, or twice per month, 24 doses. All injections will be given at the clinic.
  Arms: Omalizumab injection
Drug: Sodium Chloride (NaCl) 0.9 % — The study drug (omalizumab or placebo) will be given as a subcutaneous injection, which means an injection into the fat layer just under the skin in your arm or leg. This is similar to an insulin injection and not as deep as a typical vaccine injection. After the injection, participants will be monitored for any side effects. The study team will determine the dose and how often the injection is given based on the participant's weight and blood test results. Injections will be either be given monthly, 12 doses, or twice per month, 24 doses. All injections will be given at the clinic.
  Arms: Placebo injection

SUMMARY:
This research is being done to test if a drug called omalizumab can help people with Chronic Obstructive Pulmonary Disease (COPD) and allergies.

Each participant will be in the study for about 16 months, including 1-3 months of screening, 12 months of receiving the study drug at a clinic, and a follow-up call one month after your final clinic visit.

DETAILED DESCRIPTION:
This study is for people 40 years and older with COPD who also have allergens in their home that they are allergic to, like pet dander, cockroaches or dust mites.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent.
* Age >40 years at screening.
* Combustible tobacco cigarette exposure >10 pack-years.
* Self-report of physician diagnosis of COPD and currently on dual or triple long-acting inhaled therapy (ICS/LABA/LAMA, ICS/LABA, LABA/LAMA).
* COPD Assessment Test (CAT) score of >15 OR history of at least one documented moderate (requiring treatment with oral corticosteroids) or severe (requiring ED visit or hospitalization) COPD exacerbation in the past year.
* Participants of childbearing potential must have negative pregnancy test upon study entry.
* Female (and male) participants with reproductive potential must agree to use FDA approved methods of contraception for duration of study.
* Post-bronchodilator FEV1/FVC ratio < 0.7 and FEV1% predicted < 80%.
* Sensitization to one or more of five common indoor allergens including cat, dog, mouse, cockroach, dust mite defined with positive skin prick test (SPT) (SPT wheal size at least 3 mm greater than negative control). Positive specific IgE testing within 12 months of randomization to cat, dog, mouse, cockroach, or dust mite will be accepted in lieu of skin prick test if SPT is not interpretable or SPT cannot be safely performed.
* Exposure to the same allergen to which individual is sensitized based on measurement in home settled dust (1 U/g cockroach, 1 μg/g mouse, 2 μg/g dust mite, (Der f 1), 8 μg/g for cat and dog).

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
* Live in a location other than home (i.e., care facility)
* Actively breastfeeding.
* Current asthma diagnosis.
* Other lung disease (cystic fibrosis, pneumoconiosis, bronchiectasis or otherwise) that is considered the primary respiratory diagnosis and would interfere with participation in the study
* Reduced life expectancy due to other disease that in the opinion of the investigator may interfere with participation in the study.
* Participants with severe medical condition(s) that in the view of the investigator prohibits participation in the study.
* Received or listed for a lung transplant.
* Surgical or bronchoscopic lung volume reduction surgery in the 12 months prior to screening.
* History of infection or active infection due to Mycobacterium tuberculosis
* Active parasitic infection diagnosed and/or treated within 6 months of randomization
* Currently receiving allergen immunotherapy.
* History of anaphylaxis from medications, foods or otherwise.
* Current active prescription for epinephrine autoinjector for treatment of severe chronic urticaria.
* Known sensitivity to study drug(s) or another biologic medication.
* Use of any other investigational agent for COPD in the last 90 days. If the other investigational agent being used is a biologic agent, this must be washed out for 6 months prior to randomization.
* Active use of biologic medication (monoclonal antibody) for treatment of respiratory disease in the past 6 months (benralizumab, omalizumab, mepolizumab, resilizumab, dupliumab, tezepelumab, or other similar medication or use of biologic medication for treatment of any non-respiratory disease in the past 3 months.
* Use of chronic systemic corticosteroids at doses above 10mg daily prednisone or the equivalent.
* Use of systemic corticosteroid course for acute exacerbation of COPD within 4 weeks of randomization.
* Weight < 66 or >330 lbs; and total IgE < 30 IU/mL or >700 IU/mL; or no available dosing recommendation based on weight and total IgE level.
* No ICS in background regimen for individuals with blood eosinophil count of >300 and systemic steroid requiring exacerbation in the past year, except in case of contraindication to ICS such as thrush, osteoporosis, or pneumonia in the past year.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Rate of COPD exacerbations | 12 months
  To determine the efficacy of omalizumab injection in reducing the annualized rate of moderate or severe exacerbations (primary outcome) over the course of 12 months among individuals with COPD having sensitization and exposure to any of a panel of common indoor aeroallergens.

CONTACTS AND LOCATIONS:
Overall Officials: Nirupama Putcha, Principal Investigator — Johns Hopkins School of Medicine; Elizabeth Sugar, PhD, Principal Investigator — Johns Hopkins University
Locations (23):
- United States (23):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona- Tuscon, Tucson, Arizona
  - University of San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Florida, Jacksonville, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Mount Sinai, Icahn School of Medicine, New York, New York
  - Columbia University, New York, New York
  - Cornell University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Vermont, Colchester, Vermont
  - Pacific Northwest Airways - VA Puget Sound Healthcare System, Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No